CLINICAL TRIAL: NCT02023970
Title: TRANSLINK: A Prospective, Multi-center, Multi-national, Non Randomized, Open, Study to Defining the Role of Xeno-directed and Immune Events (SVD) in Patients Receiving Animal-derived Bioprosthetic Heart Valves.
Brief Title: TRANSLINK: Defining the Role of Xeno-directed and Immune Events (SVD) in Patients Receiving Animal-derived Bioprosthetic Heart Valves
Acronym: TRANSLINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RC13_0241
Record Dates: First submitted 2013-12-05; First posted 2013-12-30 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Patients Receiving Animal-derived Bioprosthetic Heart Valves
Keywords: Bioprosthetic heart valves, immune response, structural valve deterioration, valvular disease
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase A: Diagnostic Study (Other): Objective: to assess the differential immune response in patients with or without SVD (given the low rate of SVD) a matched cases-controls study allows a powerful statistical analysis avoiding main confounding factors for a first discovery of a SVD-specific immune response. Results will be validated in prospective Phase B.
  Interventions: Device: Patients receiving animal-derived bioprosthetic heart valves.; Other: Echocardiography (1); Biological: Blood sample (1)
- Phase B1 (Prospective Study): Cohort of prevalent patients (Other): This cohort is specifically designed to study the kinetics of the immune response before and after implantation of an aortic BHV. Eight of the most frequently implanted BHV worldwide will be assessed:
  Interventions: Device: Patients receiving animal-derived bioprosthetic heart valves.; Other: Echocardiography (2); Biological: Blood sample (2)
- Phase B2 (Prospective Study): Cohort of incident patients (Other): Due to the low incidence of SVD during the first 4 post-operative years, a second cohort will be constituted by patients undergone biological aortic valve replacement at least 5 years before. The objective of this second cohort is to cover a period of time where risk of SVD occurrence is potentially high.
  Interventions: Device: Patients receiving animal-derived bioprosthetic heart valves.; Other: Echocardiography (3); Biological: Blood sample (3)

INTERVENTIONS:
Device: Patients receiving animal-derived bioprosthetic heart valves.
Other: Echocardiography (1)
  Other Names: Echocardiography at the baseline (inclusion visit)
  Arms: Phase A: Diagnostic Study
Other: Echocardiography (2)
  Other Names: Echocardiography will be performed at visits before surgery, 6, 24 and 42 months at inclusion site.
  Arms: Phase B1 (Prospective Study): Cohort of prevalent patients
Other: Echocardiography (3)
  Other Names: At inclusion visit and:; - If normal echocardiographic parameters (without SVD signs): echocardiography at 42 months.; - If subnormal echocardiographic parameters (SVD signs): echocardiographic follow-up will be performed on site at 1 year and 42 months.
  Arms: Phase B2 (Prospective Study): Cohort of incident patients
Biological: Blood sample (1)
  Other Names: Blood sample will be collected at the time of SVD diagnosis in SVD patients and non -SVD control patients.
  Arms: Phase A: Diagnostic Study
Biological: Blood sample (2)
  Other Names: Blood samples will be harvested the day before the surgery and then at 1, 6, 12, 24 and 42 months, representing 6 samples per patient.
  Arms: Phase B1 (Prospective Study): Cohort of prevalent patients
Biological: Blood sample (3)
  Other Names: At inclusion visit and:; - If normal echocardiographic parameters (without SVD signs): blood samples at 2 year and 42 months; - If subnormal echocardiographic parameters (SVD signs): blood samples at 1 year and 42 months.
  Arms: Phase B2 (Prospective Study): Cohort of incident patients

SUMMARY:
Cardiac valve disorders are widely spread in the general population and represents the third most frequent cardiovascular illness after coronary disease and arterial hypertension. In this context, aortic valve stenosis (the central pathology in this project) is the most common form of valve disease. Cardiac valve replacement is in the vast majority of cases the first line therapy for degenerative heart-valve diseases. These are represented by mechanical and bioprosthetic valve (BHV). In the vast majority of cases, BHV are derived from animals and from a biological standpoint are classified as xenografts. BHV are severely penalised by a premature structural damage, with ultimate valve failure occurring around 10 years after surgery in 5 to 30% of cases, depending on the type of BHV used. Several factors [including dyslipidaemia, gender, valve position] may contribute to the ultimate failure of the BHV and there has been increasing evidence recently of a substantial immune reaction elicited by the implanted BHV. This immune response is still poorly understood. It may lead to adverse immune reactions and this will be thoroughly investigated by the TRANSLINK team. In this light, the TRANSLINK project aims to provide the necessary data to demonstrate beyond any reasonable doubt the central role of the anti-BHV immune response in the premature failure of BHV and to provide efficient strategies to enable safe implantation of BHV valves in currently unsuitable candidates

ELIGIBILITY:
Inclusion criteria

To be enrolled, the following criteria have to be fulfilled:

*Phase A: Diagnostic Study

Inclusion criteria for SVD-patients:

* Patient age: 18 to 85 years old at the time of surgery
* Echographic signs of SVD (Mean trans-valvular gradient ≥ 30 mm Hg AND Effective Orifice Area ≤ 1 cm2 worsen over time OR Aortic Insufficiency > grade 2/4)
* Single aortic valve replacement +/- associated to CABG, Bental, Mitral or Tricuspid repair, aortic surgery, Radiofrequency.
* First cardiac surgery (no multiple cardiac surgeries)
* No immunosuppressive regimen any time within the 6 months prior surgery.
* - No use of other allo or xenogenic tissue than aortic valve prosthesis during cardiac surgery
* Patient has been informed of the nature of the study, agrees to its provisions and has signed the informed consent form prior to any study related procedure
* Patient agrees to undergo all protocol required follow-up examinations and requirements at the investigational site

Non-SVD patients (control-patients):

* Patients will be defined as patients operated on with an aortic BHV without echographic signs of SVD and matched for: Age at surgery (±2 years), type of BHV and follow-up time (± 6 months).
* Patient has been informed of the nature of the study, agrees to its provisions and has signed the informed consent form prior to any study related procedure
* Patient agrees to undergo all protocol required follow-up examinations and requirements at the investigational site

To increase the statistical power (which cannot be calculated according to the novelty of the project), two controls will be matches with each SVD-Case.

*Phase B: Prospective Study

B1: Cohort of prevalent patients

* Patient age: 18 - 85 years old at the time of surgery
* Patient scheduled for single aortic valve replacement with a BHV (surgical or percutaneous valve) +/- associated to CABG, Bental, Mitral or Tricuspid repair, aortic surgery, Radiofrequency.
* First cardiac surgery (no multiple cardiac surgeries)
* No immunosuppressive regimen any time within the 6 months prior surgery and no immunosuppressive regimen after surgery.
* No use of other allo or xenogenic tissue than aortic valve prosthesis during cardiac surgery
* Patient is affiliated to the Social Security or equivalent system
* Patient has been informed of the nature of the study, agrees to its provisions and has signed the informed consent form prior to any study related procedure
* Patient agrees to undergo all protocol required follow-up examinations and requirements at the investigational site Eight of the most frequently implanted BHV worldwide will be assessed: 1 surgical porcine valve: Mosaic (Medtronic); 4 surgical bovine pericardium valves: Perimount-Carpentier (Edwards), Magna ease (Edwards), Trifecta (St. Jude Medical) and the Mitroflow PRT valve (Sorin); 1 surgical equine valve: 3F-valve or Enable (Medtronic) and 2 percutaneous pericardium valves (TAVI): Corevalve (porcine pericardium - Medtronic) and Sapien valve (bovine pericardium - Edwards).

Fifty patients per type of BHV will be included. When 50 patients were included in one of the eight groups, we will stop the inclusions in this group.

Additionally, a control group of heart operated patients without biological valve will be included in the study (patients operated on with a mechanical valve (n=50) or for CABG without BHV (n=50).

Control group (CABG or aortic mechanical valve)

* Patient age: >65 years old for CABG and 18-85 years old for mechanical valve replacement
* Patient operated on coronary artery bypass (for CABG group)
* Patient with valve aortic replacement following aortic valve stenosis (for mechanical valve group)
* No immunosuppressive regimen any time within the 6 months prior surgery and no immunosuppressive regimen after surgery.
* No use of other allo or xenogenic tissue than aortic valve prosthesis during cardiac surgery.

B2: Cohort of incident patients

* Patient age: 18 to 85 years old (at the time of surgery) who underwent a single isolated aortic valve replacement with a BHV +/- associated to CABG, Bental, Mitral or Tricuspid repair, aortic surgery, Radiofrequency. more than 5 years ago.
* First cardiac surgery (no multiple cardiac surgeries)
* No immunosuppressive regimen any time within the 6 months before inclusion and no immunosuppressive regimen after inclusion.
* Patient is affiliated to the Social Security or equivalent system
* Patient has been informed of the nature of the study, agrees to its provisions and has signed the informed consent form prior to any study related procedure
* Patient agrees to undergo all protocol required follow-up examinations and requirements at the investigational site

As control, patients who underwent isolated CABG (n=50) or aortic mechanical valve replacement more than 5 years ago (n=50) will be enrolled.

Control group (CABG or aortic mechanical valve)

* Patient age (at the time of surgery): > 65 years old for CABG and 18-85 years old for mechanical valve replacement
* Patient operated on coronary artery bypass (for CABG group) more than 5 years ago
* Patient with valve aortic replacement following aortic valve stenosis (for mechanical valve group) more than 5 years ago
* No immunosuppressive regimen any time within the 6 months prior inclusion and no immunosuppressive regimen after inclusion.
* No use of other allo or xenogenic tissue than aortic valve prosthesis during cardiac surgery

Exclusion criteria

Any of the following is regarded as criteria for exclusion from the study:

* Female of child bearing potential
* Severe renal insufficiency: GFR <=30 ml/min/
* Severe dyslipidemia: total cholesterol >350 mg/dl, triglycerides >750 mg/dl
* Ongoing infection (patient may be evaluated for enrolment after resolution)
* HIV infection
* Active autoimmune disease
* Multiple cardiac surgeries
* Patient with immunosuppression regimen
* Presence of any condition (medical, psychological, social, or geographical), actual or anticipated, that the Investigator feels would restrict or limit the patient's successful participation for the inclusion or duration of the study
* Presence of any severe medical condition such that the patient is not expected to survive for the planned study follow-up period.
* Patient is not able to give informed consent
* Patient under trusteeship or under guardianship
* No affiliation to a social security or equivalent system
* Patient is currently participating in an investigational drug or device study that clinically interferes with the current study endpoints

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1668 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-01-10 (Actual)

PRIMARY OUTCOMES:
Echocardiography data to assess the structural valve deterioration | 5 years
  The primary endpoint to be analyzed in the study is assessment by echocardiography of structural valve deterioration after implantation of pig valve or bovine pericardium valve or equine pericardium valve.
  TRANSLINK project aims primarily at establishing the possible role of recipient immune response against biological prosthetic heart valves as a major cause to mid-long-term structural valve deterioration and clinical dysfunction.

SECONDARY OUTCOMES:
Process of valve degeneration according to the type of BHV | 5 years
  To study the process of valve degeneration according to the type of BHV (porcine, bovine or equine BHV or type of industrial process) and BHV clinical outcome.
Large international and prospective patient's cohort and clinical database with a biocollection | 5 years
  To implement a large international and prospective patient's cohort and clinical database with a biocollection (biobank) of patients receiving an aortic BHV to identify immune biomarkers following aortic valve replacement.
Clinic-biological correlations | 5 years
  To analyse clinic-biological correlations prospectively following BHV.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-christian ROUSSEL, Professor, Study Chair — Nantes University Hospital; Gino GEROSA, Professor, Principal Investigator — University of Padova Medical School, Italy; Rafael MAÑEZ, Professor, Principal Investigator — University Hospital of Bellvitge, Barcelona, Spain; Manuel GALIÑANES, Professor, Principal Investigator — University Hospital Vall d'Hebron, Barcelona, Spain
Locations (5):
- University of Manitoba, Winnipeg, Manitoba, Canada
- Nantes University Hospital, Nantes, France
- University of Padova Medical School, Italy, Padua, Italy
- Spain (2):
  - University Hospital of Bellvitge, Barcelona, Spain, Barcelona
  - University Hospital Vall d'Hebron, Barcelona, Spain, Barcelona